CLINICAL TRIAL: NCT03788720
Title: Comparison Between Suture of the Ovary Versus no Suture After Enucleation of Ovarian Endometrioma
Brief Title: Suture of the Ovary After Enucleation of Ovarian Endometrioma
Acronym: SOAVE-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOAVE-1
Record Dates: First submitted 2018-10-11; First posted 2018-12-28 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Endometrioma
Keywords: Endometrioma; Laparoscopy; Suture; Ovary
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Surgeons who perform the surgery will be not masked for the treatment allocation.
  Evaluators (sonographers, data analyzers) will be blind for the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suture (Experimental): Women undergoing suturing of the ovarian cortex after laparoscopic enucleation of endometriomas.
  Interventions: Procedure: Suture of the ovarian cortex
- No suture (Sham Comparator): Women undergoing laparoscopic enucleation of endometriomas without subsequent suture of the ovarian cortex.
  Interventions: Procedure: No suture of the ovarian cortex

INTERVENTIONS:
Procedure: Suture of the ovarian cortex — Suture of the ovarian cortex after laparoscopic enucleation of endometriomas, using one single monofilament suture material, continuous suture technique with maximum 5 transfixion of the ovarian cortex and intracorporeal knots only (no extracorporeal knots).
  Arms: Suture
Procedure: No suture of the ovarian cortex — Laparoscopic enucleation of endometriomas without suture of the ovarian cortex
  Arms: No suture

SUMMARY:
Endometriosis is an estrogen-dependent chronic disease, characterized by the presence of ectopic endometrial-like tissue outside the uterine cavity.

According to the most updated guidelines of the European Society of Human Reproduction and Embryology (ESHRE), infertile women with endometriomas smaller than 3 cm should be addressed directly to Assisted Reproduction Technology (ART); conversely, for infertile women with endometriomas larger than 3 cm, enucleation of ovarian endometriomas could be considered in order to improve reproductive outcomes (both spontaneous and ART pregnancy rate).

To date, literature data do not allow to draw a firm conclusion about the best strategy to reduce ovarian damage during enucleation of ovarian endometriomas: in particular, investigators still lack robust evidence in order to choose between suturing the ovary or not after the enucleation.

In this scenario, the aim of our the study will be to compare functional outcomes of the ovary in a group of women undergoing suturing of the ovarian cortex after laparoscopic enucleation of endometriomas (cases) and a group of women undergoing laparoscopic enucleation of endometriomas without subsequent suture of the ovarian cortex.

ELIGIBILITY:
Inclusion Criteria:

* Women affected by one primary (no recurrent) monolateral ovarian endometrioma, with maximum diameter between 5 and 10 cm, undergoing laparoscopic enucleation by stripping technique;
* Normal AFC at the enrollment (baseline).

Exclusion Criteria:

* Any other disease;
* Bilateral endometriomas;
* Deep infiltrating endometriosis;
* No previous pelvic surgery (even not gynecological);
* Any other pharmacologic and non pharmacologic treatment in the previous 3 months (wash-out period);

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Antral Follicle Count (AFC) | Change from day 3 of the menstrual cycle prior to the elective laparoscopic surgery to day 3 of the menstrual cycle after to the elective laparoscopic surgery
  AFC will be evaluated on day 3 of the cycle by a transvaginal ultrasound. Initially the ovarian volume of both the ovaries is calculated. Further the number of small antral follicles in both the ovaries is measured. These follicles could vary in size from 2-10 mm.

SECONDARY OUTCOMES:
Pulsatility index, evaluated by Doppler flowmetry, of the ovarian artery | Change from day 3 of the menstrual cycle prior to the elective laparoscopic surgery to day 3 of the menstrual cycle after to the elective laparoscopic surgery
  Evaluation of the pulsatility index (PI; minimum: 0; maximum: 7; higher values represent a better outcome) of the ovarian artery.
Resistive index, evaluated by Doppler flowmetry, of the ovarian artery | Change from day 3 of the menstrual cycle prior to the elective laparoscopic surgery to day 3 of the menstrual cycle after to the elective laparoscopic surgery
  Evaluation of the resistive index (RI minimum: 0; maximum: 3; higher values represent a worse outcome) of the ovarian artery.
Ovarian volume | Change from day 3 of the menstrual cycle prior to the elective laparoscopic surgery to day 3 of the menstrual cycle after to the elective laparoscopic surgery
  Evaluation of the ovarian volume calculated using the prolate ellipsoid formula (length x height x width x 0.523)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Principal Investigator — Università degli Studi dell'Insubria; Fabio Ghezzi, M.D., Study Director — Università degli Studi dell'Insubria; Jvan Casarin, M.D., Principal Investigator — Università degli Studi dell'Insubria; Simone Garzon, Principal Investigator — Università degli Studi dell'Insubria
Locations (1):
- "Filippo Del Ponte" Hospital, Varese, Italy

IPD SHARING:
Plan to Share IPD: Undecided